CLINICAL TRIAL: NCT00791323
Title: Efficacy of Ketorolac 0.4% in Prostaglandin Suppression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MA-ACU-08-001
Record Dates: First submitted 2008-11-12; First posted 2008-11-14 (Estimated); Results first posted 2011-09-23 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Ketorolac; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Ketorolac 0.4%
  Interventions: Drug: Ketorolac 0.4%
- 2 (Active Comparator): Mineral Oil Emollient
  Interventions: Drug: Lubricating Eye Drop

INTERVENTIONS:
Drug: Ketorolac 0.4% — One drop 4 times a day in the pre-operative eye beginning day 0 for 4 days
  Other Names: Acular LS™
  Arms: 1
Drug: Lubricating Eye Drop — One drop 4 times a day in the operative eye beginning one day prior to the peripheral iridotomy and continuing until the day of IOL implantation
  Other Names: Soothe® XP
  Arms: 2

SUMMARY:
A pilot study to evaluate the extent of PGE2 inhibition (mean aqueous values) by Ketorolac 0.04% following peripheral iridotomy

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo phakic IOL implantation

Exclusion Criteria:

* History of intraocular surgery in the operative eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketorolac 0.4%: Ketorolac 0.4%
- Soothe® XP: Mineral Oil Emollient
Period: Overall Study
Arm/Group | Ketorolac 0.4% | Soothe® XP
Started | 6 | 3
Completed | 6 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac 0.4% | Soothe® XP | Total
Number analyzed (Participants) | 6 | 3 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 30.2 (9.7) | 33.3 (2.5) | 31.75 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Prostaglandin E2 (PGE2) Aqueous Humor Levels
Description: The mean level of PGE2 (a naturally occurring prostaglandin E2 in the eye that can cause inflammation and other complications) in the aqueous humor (the thin, watery fluid in the eye) 2 days following peripheral iridotomy (ocular surgery).
Time Frame: Day 3
Population: Intent to Treat defined as all patients who started the study (randomized) with processed aqueous samples. Two patients in the Ketorolac 0.4% arm did not have aqueous humor samples processed.
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (pg/ml)
Arm/Group | Ketorolac 0.4% | Soothe® XP
Number analyzed (Participants) | 4 | 3
Picograms per milliliter (pg/ml) | 1027.4 (429) | 1014.7 (196.8)

ADVERSE EVENTS:
Arm/Group | Ketorolac 0.4% | Soothe® XP
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo